CLINICAL TRIAL: NCT02018978
Title: Phase II RCT of Comprehensive Triaged HIV Prevention: Tanzania
Brief Title: Comprehensive Triaged HIV Prevention in Tanzania
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Muhimbili University of Health and Allied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01MH095869 (NIH)
Record Dates: First submitted 2013-12-17; First posted 2013-12-24 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: HIV
Keywords: HIV prevention; Behavioral intervention; Community-randomized trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CTHP (Experimental): 1. HIV Voluntary Counseling and Testing at Community Prevention Center-The center will be open to all community members.
  2. Community Mobilization-HIV/AIDS and VCT information will be disseminated with pamphlets, community discussions, and meetings.
  3. Risk Assessment and Triaged Counseling and Recruitment-Clients identified at high-risk for HIV infection and HIV-infected clients we be offered an additional counseling session. Participation will be incentivized. These clients will also be provided with up to 3 referral cards to give to sexual partners. If partners come for VCT, they will receive a small incentive.
  4. Incentives & Support Activities - Modest and ethically appropriate incentives, including those providing nutritional support (food), health and hygiene benefits (bed nets), transport to access interventions, or income generation potential, will be provided for participation in some project interventions, and these will be graduated based on HIV risk potential.
  Interventions: Behavioral: Comprehensive Triaged HIV Prevention (CTHP)
- Standard of Care (No Intervention): This arm will receive standard of care HIV-related services, including clinic-based voluntary counseling and testing and referrals to HIV care and treatment government-run facilities.

INTERVENTIONS:
Behavioral: Comprehensive Triaged HIV Prevention (CTHP) — 1. HIV Voluntary Counseling and Testing at Community Prevention Center-The center will be open to all community members.
  2. Community Mobilization-HIV/AIDS and VCT information will be disseminated with pamphlets, community discussions, and meetings.
  3. Risk Assessment and Triaged Counseling and Recruitment-Clients identified at high-risk for HIV infection and HIV-infected clients we be offered an additional counseling session. Participation will be incentivized. These clients will also be provided with up to 3 referral cards to give to sexual partners. If partners come for VCT, they will receive a small incentive.
  4. Incentives & Support Activities - Modest and ethically appropriate incentives, including those providing nutritional support (food), health and hygiene benefits (bed nets), transport to access interventions, or income generation potential, will be provided for participation in some project interventions, and these will be graduated based on HIV risk potential.
  Arms: CTHP

SUMMARY:
This is a 3-year Phase II trial of a HIV prevention strategy designed to significantly reduce population-level HIV incidence. The study design is a two-arm community randomized controlled trial of Comprehensive Triaged HIV Prevention (CTHP) which includes: (a) Access to an HIV center which will provide free HIV testing and counseling, (b) Educational activities related to HIV risk behavior, (c) Special counseling sessions for HIV-infected clients, (d) A onetime provision of a small amount of food or health products for sex partners of persons testing positive for HIV or reporting HIV risk behaviors when they come to receive HIV testing, (e) A post test support club for persons infected with HIV, (f) An income generation training program for people testing positive for HIV, (g) Transportation assistance in visiting the HIV Care and Treatment Clinic in the area for those who test positive for HIV, and, (h) Counseling and transportation support for those on medical treatment for HIV to assist them in attending scheduled appointments, and receiving and taking their medications as recommended by the clinic staff. The study will take place within two communities located in Kisarawe district, Tanzania. The intervention will occur over an 18-month period with outcomes assessed at baseline and post-intervention. The study hypothesis is that individuals in the intervention community will have a lower incidence of sexually transmitted infections (STIs) than those in the control community.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18-55 years of age
* Lives in the household regularly
* Able to provide informed consent
* Plans on living in the study area for the duration of the study (2 years)

Exclusion Criteria:

* Younger than 18 years of age or older than 55 years of age
* Does not reside in the household regularly
* Is not able to provide informed consent
* Does not plan on living in the study area for study duration (2 years)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 739 (Actual)
Dates: Start 2013-10; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
STI Incidence | 18 months
  Incidence of sexually transmitted infections (STI) defined as any incident case of syphilis, HIV, or herpes simplex virus-2.

SECONDARY OUTCOMES:
Safety and acceptability | 18 months (during intervention)
  Safety and acceptability of the intervention will be assessed through weekly reports detailing any adverse social or physical events related to participation in the intervention compiled by study staff.
Sexual risk behavior | 18 months
  Sexual risk behavior will be measured by assessing condom use at last sex with each sexual partner, frequency of condom use in the last 6 months with each sexual partner, and number of sexual partners in the last 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Sweat, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Muhimbili University of Health and Allied Sciences, Dar es Salaam, Tanzania